CLINICAL TRIAL: NCT01341444
Title: The Use of the Prevena Incision Management System on Closed Recipient Site Incisions in Renal Transplant Subjects
Brief Title: The Use of the Prevena Incision Management System (PIMS) on Closed Incisions in Renal Transplant Subjects
Acronym: PIMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment Difficulties
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHS.2012.Prevena.Cooper.01
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Surgical Site Reaction
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena Incision Management System (Experimental): Negative Pressure Therapy Device
  Interventions: Device: Prevena Incision Management System
- Standard of Care for Surgical Incisions (Placebo Comparator): Sterile gauze and a non-penetrable barrier
  Interventions: Other: Standard of Care for Surgical Incisions

INTERVENTIONS:
Device: Prevena Incision Management System — It is intended to manage the environment of surgical incisions that continue to drain following sutured or stapled closure by maintaining a closed environment and removing exudate via the application of negative pressure wound therapy (NPWT).
  Arms: Prevena Incision Management System
Other: Standard of Care for Surgical Incisions — Sterile 4X4 Non-Penetrable barrier
  Arms: Standard of Care for Surgical Incisions

SUMMARY:
This study is being conducted to see how safe and effective the Prevena Incision Management System "Prevena" is when placed over a renal transplantation incision. Prevena provides negative pressure (suction) wound therapy. Prevena will be tested while applied during the time each subject is hospitalized and up to 5 days after the surgery. Prevena is a small portable negative pressure device which consists of a therapy unit that delivers negative pressure. It also includes a dressing system that is intended for use over closed incisions after surgery.

The intent of this study is to evaluate Prevena versus the standard care that a doctor would use normally after a kidney transplant.

DETAILED DESCRIPTION:
This is a randomized, single-center, comparative interventional study looking at the effect of Prevena™ on renal transplant surgical Subjects compared to a control arm treated with the standard-of-care wound dressing. The prospective, post-marketing clinical study described in this protocol will assess the effectiveness and functional performance of PrevenaTM in this clinical indication.

ELIGIBILITY:
Pre-operative Inclusion Criteria

The Subject:

1. is an adult ≥ 18 years old of either gender
2. is able to provide their own informed consent Protocol: AHS.2012.Prevena.Cooper.01 v 4.0 Confidential/Property of KCI USA, Inc. Page 6 of 71
3. will undergo open renal transplant surgery within the next 30 days
4. will require a surgical incision able to be covered completely by the PIMS dressing
5. is pre-operatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class I (Clean): An uninfected operative wound in which no inflammation is encountered and the respiratory, alimentary, genital, or uninfected urinary tract is not entered

      - OR -
   2. Class II (Clean Contaminated): An operative wound in which the respiratory, alimentary, genital, or uninfected urinary tract are entered under controlled conditions and without unusual contamination
6. is willing and able to return for all scheduled and required study visits
7. if female, must test negative on serum pregnancy test
8. if a female of child-bearing potential, must be willing to utilize an acceptable method of birth control (e.g., birth control pills, condom with spermicide, diaphragm with spermicide, implants, IUD, injections, vaginal rings, hormonal skin patch, etc.) for the duration of study participation
9. is not concurrently enrolled in a clinical trial which may impact subject health or the surgical incision site

Intra-operative Inclusion Criteria Subjects must meet the following intra-operative inclusion criteria to be eligible for randomization.

The Subject:

1. continues to meet all pre-operative inclusion criteria
2. has undergone a Class I or II CDC Wound Classification procedure resulting in a closed surgical incision able to be covered completely by the PIMS dressing

Pre-operative Exclusion Criteria

The Subject:

1. has a BMI < 18.5 kg/m2 and > 40 kg/m2
2. has a systemic infection at the time of open renal transplant surgery
3. has a remote-site skin infection at the time of open renal transplant surgery
4. is preoperatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

      - OR -
   2. Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera
5. has a known allergy or hypersensitivity to silver, or drape materials that contain acrylic adhesives

Intra-Operative Exclusion Criteria Subjects who meet any of the following intra-operative exclusion criteria are considered screen failures and are not eligible for randomization.

The Subject:

1. is found to meet any of the pre-operative exclusion criteria
2. has obvious contamination of the surgical incision
3. requires external surgical drains that will be covered by the PIMS dressing
4. is determined to have a CDC Wound Classification of:

   1. Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

      - OR -
   2. Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera Protocol: AHS.2012.Prevena.Cooper.01 v 4.0 Confidential/Property of KCI USA, Inc. Page 8 of 71
5. requires a transfusion, has disseminated-intravascular coagulopathy (DIC) or other medical or surgical conditions during open renal transplant surgery deemed by the Investigator to pose a prohibitively high risk for surgical re-exploration
6. is deemed unable to continue in the study by the Investigator as the Subject's safety or well-being may be jeopardized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cooper, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena Incision Management System | Standard of Care for Surgical Incisions
Started | 31 | 32
Completed | 26 | 29
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena Incision Management System | Standard of Care for Surgical Incisions | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.71 (11.29) | 51.75 (12.19) | 50.25 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 22 | 19 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 14 | 32
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Complications (SSCs)
Description: The primary objective to compare short-term surgical incision-related clinical outcomes in Subjects undergoing open renal transplant surgery when treated with Prevena vs. the standard-of-care wound dressing. Clinical outcomes of interest are defined as Surgical Site Complications (SSCs) that include incisional fluid accumulation (i.e. seroma, hematoma, abscess), dehiscence, surgical site infection (SSI). These outcomes will be compared to a control group consisting of subjects screened for the same inclusion/exclusion criteria but treated with standard-of-care incision dressing.
Time Frame: 62 Days
Population: Analysis of this endpoint was based on the Full analysis Set (FAS population). The FAS population consists of participants who met all of the pre- and intra-operative eligibility criteria, were randomized and received treatment. Subjects without SSC must have received 5 days of Prevena or at least 3 days of SOC dressing and completed 30 day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena Incision Management System | Standard of Care for Surgical Incisions
Number analyzed (Participants) | 28 | 30
Participants | 6 | 8

ADVERSE EVENTS:
Arm/Group | Prevena Incision Management System | Standard of Care for Surgical Incisions
Serious Adverse Events (participants affected / at risk) | 11/31 | 13/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevena Incision Management System (N=31) | Standard of Care for Surgical Incisions (N=32)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Kidney Transplant Rejection (Immune system disorders) | 2 | 0
Wound Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Blood Creatine Increased (Investigations) | 1 | 1
Urine Output Decreased (Investigations) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular (Nervous system disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Incisional Drainage (Surgical and medical procedures) | 0 | 1
Ebolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No